CLINICAL TRIAL: NCT06301477
Title: PRecisiOn Microbiome Directed ExtensiOn of Anti-TNFα Crohn's Disease ThErapy in Children: The PROMOTE Trial
Acronym: PROMOTE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, David Mack, Director, CHEO IBD Centre, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 23/109X
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
Keywords: Resistant Starch; Microbiome; anti-TNF
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, placebo-controlled, double-blinded, pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treating physician, study participants, and research coordinators and lab researchers will not have knowledge of the randomization codes and will be blinded as to study product allocation. Unblinding will occur only if necessary to ensure study participants safety. Only Dr. Mack (Co-PI) will request to break the blind for safety reasons. Once the blind is broken by Dr. Mack the patient will be discontinued from study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch (Active Comparator): Once daily oral consumption of either 7.5g/m2 or 5.0g/m2 (body surface area) of a resistant starch for 48 weeks that is individually optimized at 24 weeks.
  Interventions: Other: Resistant Starch
- Placebo (Placebo Comparator): Once daily oral consumption of a readily digestible food-grade cornstarch that resembles the study product in appearance, smell and taste for 48 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Resistant Starch — 7.5g/m2 or 5.0g/m2 (body surface area) resistant starch oral consumption
  Arms: Resistant Starch
Other: Placebo — Placebo oral consumption of food-grade cornstarch
  Arms: Placebo

SUMMARY:
To determine whether a specific food-origin plant-derived resistant starch (RS) optimized for the individual will increase the abundance of known butyrate producing microbes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8.0 to 16.9 years of age.
* Capable of giving informed consent, or if appropriate, have an acceptable representative capable of giving consent on the participant's behalf.
* Established Crohn's Disease (CD) diagnosis with the site of disease involving at least the terminal ileum or ascending colon.
* CD is in clinical remission or with mild stable disease activity (weighted Pediatric Crohn's Disease Activity Index of 0 to 39.5).
* Receiving infliximab or adalimumab anti-TNFa monoclonal antibody medication for treatment of CD.
* No changes in medical treatment for the previous month and without anticipated changes for the next month.
* Ability and willingness to comply with study procedures (e.g., stool collection) for the entire length of the study.

Exclusion Criteria:

* Allergy to RS or excipients.
* Co-existing diagnosis with diabetes mellitus type 1.
* Treatment with another investigational drug or intervention throughout the study.
* Current illicit drug or alcohol dependence.
* Inability or unwillingness of an individual or legal guardian to give written informed consent.
* Other conditions requiring immunomodulating or biological medications.
* Pregnancy.
* Participant's microbiota does not increase butyrate production utilizing any RS from the assembled panel as measured through the RapidAIM ex vivo assay.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Measure of butyrate production by assessing expression of enzymes using metaproteomic/transcriptomic analysis | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks.
  Measures of restoration and sustainment of butyrate production by using metaproteomic/transcription to assess the expression of enzymes invovled in butyrate production
Measure of butyrate production by assessing production of shorty-chain-fatty-acids including butyrates using metabolomics analysis | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks.
  Measures of restoration and sustainment of butyrate production by using metabolomics analysis to assess production of short-chain-fatty acids including butyrate.
Measure of butyrate production by assessing increases in butyrate producers using metagenomics/16S analysis | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks.
  Measures of restoration and sustainment of butyrate production by metagenomics/16s analysis to assess increases in butyrate producers

SECONDARY OUTCOMES:
Change in intensification as measured by anti-TNFa dose escalation | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  To help contextualize the anti-TNFa dose escalation (if applicable), Infliximab or adalimumab information will be recorded at baseline, 12 weeks, 24 weeks, 36 weeks and 48 weeks after start of study product. Type of anti-TNFa drug prescribed, amount of anti-TNFa prescribed, dose changes in timing of administration, trough drug serum levels, weight changes and reason for dose changes will be recorded
Change in intensification as measured by anti-TNFa interval shortening | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  To help contextualize the anti-TNFa interval shortening (if applicable), Infliximab or adalimumab information will be recorded at baseline, 12 weeks, 24 weeks, 36 weeks and 48 weeks after start of study product. Type of anti-TNFa drug prescribed, amount of anti-TNFa prescribed, dose changes in timing of administration, trough drug serum levels, weight changes and reason for dose changes will be recorded
Change in disease activity | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Weighted Pediatric Crohn's Disease Activity Index (wPCDAI) ranges from 0 to 125 points (<12.5 = remission, 12.5 to 40.0 = mild, >40.0 = moderate, >57.5 = severe).
Changes in intestinal mucosal inflammation by measuring fecal calprotectin through stool samples | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Measure of fecal calprotectin
Changes in biomarkers of inflammation by measuring c-reactive protein through blood samples | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Measure of c-reactive protein
Changes in patient reported disability outcomes as measured by the IBD Disability Index Questionnaire | Baseline, 24 weeks, 48 weeks
  The IBD Disability Index consists of 28 questions and a higher overall score is indicative of greater disability.
Changes in patient reported quality of life outcomes as measured by the IMPACT III Questionnaire | Baseline, 24 weeks, 48 weeks
  The IMPACT III questionnaire ( a health related quality of life questionnaire) consists of 35 questions and ranges in score from 0 to 231. A higher score represents a higher quality of life.
Changes in parent/caregiver reported quality of life outcomes as measured by the IMPACT III-P | Baseline, 24 weeks, 48 weeks
  The IMPACT III-P questionnaire ( a health related quality of life questionnaire) consists of 35 questions and ranges in score from 0 to 231. A higher score represents a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No